CLINICAL TRIAL: NCT05873647
Title: Effect of Inhaled Nitric Oxide on Pulmonary Ventilation/Perfusion Ratio Assessed by Electrical Impedance Tomography in Patients With Acute Respiratory Distress Syndrome
Brief Title: Effect of Inhaled Nitric Oxide on Pulmonary Ventilation/Perfusion Ratio Assessed by EIT in Patients With ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, XiaoJing Zou,MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: INOEIT20230404
Record Dates: First submitted 2023-05-10; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Electrical impedance tomography was used to monitor changes in pulmonary perfusion distribution and V/Q ratio before and after iNO in patients with acute respiratory distress syndrome to investigate the factors predicting iNO reactivity and the physiological mechanism underlying changes in oxygenation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years;
2. Patients are intubated and mechanically ventilated.

Exclusion Criteria:

1. EIT contraindications such as chest wound dressing, pacemaker installation, defibrillator, etc;
2. With a history of cerebral hemorrhage in the past half year, as well as bleeding in any site of the body;
3. Pneumothorax;
4. Medium or massive pleural effusion;
5. Refractory shock;
6. Pregnant
7. With chronic kidney disease
8. Atrial fibrillation or other malignant arrhythmia leads to a decrease in cardiac output;
9. Failure to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Lung ventilation/perfusion ration | 3 hours
  Lung ventilation/perfusion ration after iNO assessed by EIT

SECONDARY OUTCOMES:
Lung perfusion distribution | 30minutes and 3 hours
  Lung ventilation/perfusion ration after iNO assessed by EIT
Shunting | 30minutes and 3 hours
  Lung shunting% after iNO assessed by EIT
Dead space | 30minutes and 3 hours
  Lung dead space after iNO assessed by EIT
Oxygenation index | 30minutes and 3 hours
  Oxygenation index= arterial partial pressure of oxygen/fraction of inspired oxygen
Arterial partial pressure of carbon dioxide (PaCO2) | 30minutes and 3 hours
  PaCO2 is one of the key indicators of pulmonary ventilation which can be obtained from arterial blood gas analysis.
Static respiratory compliance (Crs) | 30minutes and 3 hours
  Crs=tidal volume/driving pressure
Cardiac output | 30minutes and 3 hours
  Cardiac output assessed by echocardiography
Right ventricular function | 30minutes and 3 hours
  Right ventricular function assessed by echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Hongling Zhang, Wuhan, Hubei, China